CLINICAL TRIAL: NCT06738914
Title: Twenty Years of Pancreatic Surgery in Iceland: a Retrospective Cohort Study
Brief Title: Twenty Years of Pancreatic Surgery in Iceland
Status: Completed | Type: Observational
Sponsor: Linkoeping University (Other Government)
Collaborators: Landspitali University Hospital (Other)
Responsible Party: Principal Investigator, Karin Johansen, MD, PhD, Principal investigator, Linkoeping University
Other Study IDs: VSN-24-124
Record Dates: First submitted 2024-12-12; First posted 2024-12-18 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Pancreatectomy; Pancreatoduodenectomy; Distal Pancreatectomy (DP)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A retrospective analysis of patients undergoing pancreatic operations in Landspitali University Hospital, Reykjavik, Iceland, between 2003 and 2022.

ELIGIBILITY:
Inclusion Criteria:

* All patients who have undergone pancreatic resection in Iceland between 2003-2022.
* For the secondary outcome of duodenal cancer, patients with duodenal cancer who did not undergo resection in the same time span will also be included.

Exclusion Criteria: None.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who have undergone pancreatic resection in Iceland between 2003-2022. For the secondary outcome of duodenal cancer, patients with duodenal cancer who did not undergo resection in the same time span will also be included.
Sampling Method: Non-Probability Sample
Enrollment: 244 (Actual)
Dates: Start 2003-01 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Severe complications | 2003-2022
Short-term mortality | 2003-2022

SECONDARY OUTCOMES:
Demographic, operative and postoperative data | 2003-2022
Oncological data and survival among patients with pancreatic and periampullary cancer | 2003-2022
Outcomes after pancreatic surgery among patients who underwent resection for cystic lesions | 2003-2022
Comparison of patients who underwent minimally invasive distal pancreatectomy during the study period to those who underwent open distal resection. | 2003-2022
Demographic and histopathological data as well as survival compared between patients with duodenal cancer who underwent resection and patients who did not. | 2003-2022
Trends over time in the usage of pancreatic and minimally invasive surgery as well as changes in outcomes. | 2003-2022

IPD SHARING:
Plan to Share IPD: No
Not included in the ethical approval for the study.

REFERENCES:
- [Derived] Johansen K, Birgisson G, Haraldsdottir KH. Early implementation of laparoscopic left-sided pancreatectomy in a tertiary low-volume hospital. Scand J Surg. 2025 Sep;114(3):334-341. doi: 10.1177/14574969251343471. Epub 2025 May 26. PMID 40417843

DOCUMENTS (1):
  • Study Protocol (2023-07-16): https://cdn.clinicaltrials.gov/large-docs/14/NCT06738914/Prot_000.pdf